CLINICAL TRIAL: NCT04667195
Title: Clinical Characteristics of Acutely Hospitalized Adults With Acute Pyelonephritis in the Emergency Department: A Cross-sectional Study
Brief Title: Clinical Characteristics of Acutely Hospitalized Adults With Acute Pyelonephritis
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-12a-2020
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Acute Pyelonephritis
Keywords: symptoms; Acute Pyelonephritis; clinical characteristics; upper urinary tract infection; Emergency department
MeSH Terms: conditions — Urinary Tract Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected acute pyelonephritis: Diagnosis of APN suspected at the initial clinical assessment by the receiving emergency department physician
  Interventions: Other: Clinical assessment

INTERVENTIONS:
Other: Clinical assessment — Within 4 hours of admission to the emergency department, clinical assessment will include:
  * Demographics,
  * comorbidity,
  * symptoms,
  * objective findings,
  * triage at admission,
  * blood test results,
  * urine test results

SUMMARY:
Acute pyelonephritis is an acute infection. Today the diagnosis is made primarily on the basis of unspecific clinical symptoms with flank tenderness combined with as a key clue. This study will investigate which clinical and paraclinical characteristics available within 4 hours of hospital stay, that describes the patients admitted in the emergency department with acute pyelonephritis the best.

DETAILED DESCRIPTION:
Acute pyelonephritis (APN) is a severe acute infection in the upper urinary tract, which quite frequently is seen in the emergency department (ED). In our study, we define APN as a urinary tract infection with extension above the bladder, implicated by systemic affection in a suspected urinary tract infection (ie, fever, chills, malaise and/or lethargy beyond normal, signs of sepsis). Most often, an infection of the bladder ascends to the kidneys, causing APN. Symptoms and clinical affection range from mild to severe, but it is always important to recognize and treat APN fast in order to prevent progression to sepsis, renal failure and ultimately death.

The diagnosis APN is primarily made clinically based on symptoms and supported by elevated biomarkers such as C-reactive protein (CRP) and leucocytes, and positive urinary test strips. The diagnostic process can be challenging as there is often weak and atypical symptoms.

The classic symptoms indicating APN is flank tenderness, fever and nausea/vomiting. Typical symptoms of cystitis (dysuria, pollakisuria, suprapubic pain, hematuria) are possible but often absent. Especially elderly can present with more generalized signs of infection with nothing clearly indicating localization to the urinary tract. A positive urine culture verifies the diagnosis, but it is only available after a minimum of 24 hours.

In this study, we seek to identify and quantify the patient characteristics available within 4 hours of hospital stay in patients with APN. The objectives are:

* To identify clinical and paraclinical relevant information available within 4 hours of admission that are associated with APN patients
* To investigate the association between adverse events and clinical and paraclinical relevant information in patients with APN.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of APN assessed by the receiving physician.

Exclusion Criteria:

* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely admitted patients with suspected APN from three emergency departments in the Region of Southern Denmark (Hospital Sønderjylland, Hospital Lillebælt, Odense University Hospital)
Sampling Method: Probability Sample
Enrollment: 966 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Verified and non verified APN | 2 months after patient discharge
  The decision of whether patients admitted with suspicion of APN actually has a final diagnosis of APN is based on a combination of all findings during admission. The verification of diagnosis requires human handling, interpretation and judgment. Therefore, in this study, an expert panel will define the reference standard for the diagnosis APN. The expert panel consists of two independent consultants from the emergency department with significant experience in emergency medicine and acute infections. They will individually determine whether or not the patient admitted suspected with APN actually had this diagnosis. The final diagnosis will be based on all available relevant information from the patient medical record including MRI of the kidneys. A standardized template will be used. Disagreement will be discussed until a consensus is reached.

SECONDARY OUTCOMES:
Intensive care treatment | within 60 days from admission to the emergency department
  Transfer to the intensive care unit will be recorded during the current hospitalization as a binary variable (transferred/not-transferred)
Length of hospital stay | within 60 days from current admission to the emergency department
  days spent in hospital during current admission
30-days mortality | within 30 days from arrival day
  binary
Readmission | 30 days from day of discharge
  If a subject is admitted over a 30 day period after the current hospitalization discharge measured as a binary outcome
In-hospital mortality | within 60 days from current admission to the emergency department
  binary

OTHER OUTCOMES:
90-days mortality | within 90 days from day of admission
  binary
Level of infection markers | within 4 hours from admission
  Concentration of serum procalcitonin, CRP and suPAR
Urological intervention | within 60 days from current admission to the emergency department
  Binary
Bacteriuria | within 4 hours from admission
  Binary outcome defined by microbiologist on urine culture analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Study Chair — Institute for Regional Health Research
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson JR, Russo TA. Acute Pyelonephritis in Adults. N Engl J Med. 2018 Jan 4;378(1):48-59. doi: 10.1056/nejmcp1702758. No abstract available. PMID 29298155
- [Background] Ramakrishnan K, Scheid DC. Diagnosis and management of acute pyelonephritis in adults. Am Fam Physician. 2005 Mar 1;71(5):933-42. PMID 15768623
- [Derived] Skjot-Arkil H, Cartuliares MB, Heltborg A, Lorentzen MH, Hertz MA, Kaldan F, Specht JJ, Graumann O, Lindberg MJH, Mikkelsen PA, Nielsen SL, Jensen J, Roge BT, Rosenvinge FS, Mogensen CB. Clinical characteristics and diagnostic accuracy of preliminary diagnoses in adults with infections in Danish emergency departments: a multicentre combined cross-sectional and diagnostic study. BMJ Open. 2024 Dec 5;14(12):e090259. doi: 10.1136/bmjopen-2024-090259. PMID 39638587
- [Derived] Skjot-Arkil H, Heltborg A, Lorentzen MH, Cartuliares MB, Hertz MA, Graumann O, Rosenvinge FS, Petersen ERB, Ostergaard C, Laursen CB, Skovsted TA, Posth S, Chen M, Mogensen CB. Improved diagnostics of infectious diseases in emergency departments: a protocol of a multifaceted multicentre diagnostic study. BMJ Open. 2021 Sep 30;11(9):e049606. doi: 10.1136/bmjopen-2021-049606. PMID 34593497